CLINICAL TRIAL: NCT03338920
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of ONZETRA® Xsail® (Sumatriptan Nasal Powder) for the Acute Treatment of Episodic Migraine With or Without Aura in Adolescents
Brief Title: Study to Assess the Safety and Efficacy of ONZETRA® Xsail® for the Acute Treatment of Episodic Migraine With or Without Aura in Adolescents
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: eDiary data collected not sufficient to utilize in the analysis of protocol endpoints
Sponsor: Currax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-AVP-825-301
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-06

CONDITIONS: Acute Migraine With or Without Aura
Keywords: acute migraine; aura; sumatriptan nasal powder; AVP-825; adolescents
MeSH Terms: conditions — Epilepsy | interventions — Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sumatriptan nasal powder (Experimental): Participants will be dosed with 22 milligrams (mg) sumatriptan nasal powder via two nosepieces (11 mg per nosepiece).
  Interventions: Drug: sumatriptan nasal powder
- Placebo (Placebo Comparator): Participants will be dosed with matching placebo via nosepieces containing capsules filled with lactose instead of sumatriptan.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sumatriptan nasal powder — nasal powder administered via nosepiece
  Other Names: AVP-825; ONZETRA® Xsail®
  Arms: Sumatriptan nasal powder
Drug: Placebo — lactose monohydrate powder administered via nosepiece
  Arms: Placebo

SUMMARY:
This study will be conducted to evaluate the safety and efficacy of sumatriptan nasal powder (AVP-825) compared to placebo in the acute treatment of migraine in adolescent participants, 12 through 17 years of age.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study evaluating AVP-825 for the acute treatment of migraine with or without aura in adolescent subjects (12 to 17 years old).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 12 to 17 years (inclusive) of age at the time of informed consent
* Have a diagnosis of episodic migraine with or without aura according to International Classification of Headache Disorders-Third edition, beta version (ICHD-IIIB, 1.2.1 or 1.1) criteria, for at least 1 year prior to the screening/enrollment visit
* Experienced migraine attacks of moderate-to-severe intensity and typically lasting ≥ 3 hours untreated, occurring at a frequency of ≥ 2 to ≤ 14 attacks per month for the past 6 months prior to the screening/enrollment visit
* Participant's parent or legal guardian must be willing to sign a copy of the informed consent form as well as documentation for Written Authorization for Use and Release of Health and Research Study Information, after the nature and risks of study participation have been fully explained. Participants must be willing to provide informed assent.

Exclusion Criteria:

* Participants with ≥ 15 headache days per month in total (migraine, probable migraine, or tension-type)
* Participants with the following headache types: retinal (ICHD-IIIB, 1.2.4), with brainstem aura (ICHD-IIIB, 1.2.2), hemiplegic (ICHD-IIIB, 1.2.3), status migrainosus (ICHD-IIIB, 1.4.1), other forms of complicated migraine, or secondary headaches
* Participants who have not responded to an adequate dose and appropriate duration of treatment with 2 or more triptans
* Participants with known nasal obstruction, current uncontrolled nasopharyngeal illness, or known velum insufficiency (i.e., a cleft palate and/or structural abnormalities in the soft palate and nasopharynx) that may interfere with the proper use of study medication
* Participants whose conditions in the investigator's opinion may put the participant at significant safety risk or confound the study results. This includes participants who in the investigator's opinion should not be enrolled in the study due to the risks described in the Warnings and Precautions or Contraindications sections of the ONZETRA Xsail Prescribing Information.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kyle, MD, Study Chair — Currax Pharmaceuticals
Locations (39):
- United States (39):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Advanced Research Center, Anaheim, California
  - Axis Clinical Trial Network, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Alpine Clinical Research Center, Inc., Boulder, Colorado
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - New England Institute for Neurology and Headache, Stamford, Connecticut
  - International Research Partners, LLC, Doral, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Eastern Research, Inc., Hialeah, Florida
  - South Florida Clinical Trials, Hialeah, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Clinical Integrative Research Center of Atlanta, Atlanta, Georgia
  - St. Luke's Health System, Meridian, Idaho
  - AMITA Health Medical Group Pediatric Neurology, Hoffman Estates, Illinois
  - UK Headache Center Kentucky Neuroscience Institute, Lexington, Kentucky
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Center for Pharmaceutical Research, LLC, Kansas City, Missouri
  - Clinvest Research, LLC., Springfield, Missouri
  - Meridian Clinical Research, LLC, Hastings, Nebraska
  - Meridian Clinical Research, LLC, Lincoln, Nebraska
  - Bio Behavioral Health, Toms River, New Jersey
  - Dent Neurosciences Research Center, Amherst, New York
  - New York Clinical Trials, Brooklyn, New York
  - NYCT, A Member of the Alliance, Inc., New York, New York
  - Headache Wellness Center, Greensboro, North Carolina
  - Hometown Urgent Care and Research, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - Lynn Health Science Institute, Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Road Runner Research, San Antonio, Texas
  - Olympus Family Medicine, Salt Lake City, Utah
  - South Ogden Family Medicine/CCT Research, South Ogden, Utah
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sumatriptan Nasal Powder | Placebo
Started | 79 | 80
Completed | 75 | 74
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sumatriptan Nasal Powder | Placebo | Total
Number analyzed (Participants) | 79 | 80 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 79 | 80 | 159
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 14.4 [12 to 17] | 14.4 [12 to 17] | 14.4 [12 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 42 | 90
  Male | 31 | 38 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 63 | 120
  Not Hispanic or Latino | 22 | 17 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 64 | 69 | 133
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 79 | 80 | 159

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Headache Pain Free at 120 Minutes After Treatment
Description: Participants will self-report the severity of their headache.
Time Frame: 120 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Sumatriptan Nasal Powder | Placebo
Number analyzed (Participants) | 79 | 80
Participants | 8 | 9

ADVERSE EVENTS:
Time Frame: up to approximately 28 weeks
Arm/Group | Sumatriptan Nasal Powder | Placebo
All-Cause Mortality (participants affected / at risk) | 3/79 | 2/80
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/80
Other Adverse Events (participants affected / at risk) | 3/79 | 2/80
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sumatriptan Nasal Powder (N=79) | Placebo (N=80)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT03338920/Prot_SAP_000.pdf